CLINICAL TRIAL: NCT03939390
Title: Conventional Stimulation in Follicular Phase vs. Luteal Phase Stimulation in Patients With Suboptimal Response. Randomized Clinical Trial. SUBLUTEAL Study
Brief Title: Follicular Phase Stimulation vs. Luteal Phase Stimulation in Patients Diagnosed With Suboptimal Response
Acronym: SUBLUTEAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Jorge Sunol Sala, Dr, Instituto Bernabeu
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IB-0319-001
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Improving Ovarian Stimulation; Suboptimal Responders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- follicular phase stimulation (No Intervention)
- luteal phase stimulation (Experimental)
  Interventions: Drug: time of administration of Corifollitropin Alfa

INTERVENTIONS:
Drug: time of administration of Corifollitropin Alfa — The treatment will be identical in both arms. The difference between the arms is the moment of the Administration of Corifollitropin Alfa: follicular phase of the menstrual cycle (control group) vs. luteal phase of the menstrual cycle (study group).
  Arms: luteal phase stimulation

SUMMARY:
This study aims to investigate the difference in the number of oocytes obtained by performing ovarian stimulation in follicular phase vs. luteal phase in a population of patients with previous suboptimal response.

This is a controlled randomized clinical study.

We aim to include 41 patients diagnosed with suboptimal response who will undergo an ovarian stimulation in order to vitrify and accumulate oocytes.

The main variable for evaluating the efficacy in this exploratory study will be the number of oocyte cumulus complexes obtained.

ELIGIBILITY:
Inclusion Criteria:

* Meets Bologna criteria to be diagnosed as poor responder
* Less than 10 oocytes obtained in a prior controlled protocol of conventional ovarian stimulation
* Age < 41 years
* Body Mass Index (BMI) between 18 and 32 kg/m2
* Regular menstrual cycles between 21 and 35 days.
* Indication for in vitro fertilization
* Indication to start stimulation with 150mcg of corifollitropin alpha
* Presence of both ovaries
* Ability to participate and comply with study protocol
* Signing an informed consent form

Exclusion Criteria:

* Presence of follicles larger than 10 mm in the randomization visit
* Endometriosis stage III/IV
* Patients with less than 4 oocytes in previous ovarian stimulation and poor ovarian reserve parameters (as per Bologna criteria)
* Concurrent participation in another study

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
number of oocytes | at the end of stimulation
  number of oocytes after ovarian stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sunol J, Castillo JC, Ortiz JA, Ten J, Fuentes A, Moliner B, Martinez M, Llacer J, Guerrero J, Pitas A, Bernabeu A, Bernabeu R. Conventional follicular-phase ovarian stimulation vs. luteal-phase stimulation in suboptimal responders: a randomized controlled trial. F S Rep. 2023 Jul 27;4(4):344-352. doi: 10.1016/j.xfre.2023.07.003. eCollection 2023 Dec. PMID 38204945